CLINICAL TRIAL: NCT03718000
Title: Daily Self-weighing and Holiday-associated Weight Gain in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Associate Professor and Graduate Coordinator, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00004735
Record Dates: First submitted 2018-10-17; First posted 2018-10-24 (Actual); Results first posted 2019-06-13 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: Holiday weight gain; Daily self-weighing; Weight maintenance; Caloric titration method; Obesity; Overweight; Holiday season
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): Participants in this group received no intervention during t he holiday season
- Daily Self-Weighing (DSW) (Experimental): Participants in this group performed daily self-weighing using digital WiFi scales during the holiday season
  Interventions: Device: Daily self-weighing (DSW)

INTERVENTIONS:
Device: Daily self-weighing (DSW) — DSW was conducted using digital WiFi scales during the holiday season. Participants received electronic graphic feedback of their weight fluctuations immediately after weight measurement.
  Other Names: DSW
  Arms: Daily Self-Weighing (DSW)

SUMMARY:
Background: Previous studies report 0.4-1.5kg of weight gain during the holiday season, which may contribute to annual weight gain.

Purpose: To test whether daily self-weighing (DSW) can prevent holiday weight gain.

Hypothesis: We hypothesized that daily self-weighing would effectively prevent weight and fat gain, and that individuals with overweight and obesity would respond most favorably to DSW.

DETAILED DESCRIPTION:
A single-blinded randomized control trial:

Adults (age 18-75y, BMI ≥ 18.5kg/m2) were randomized to either a control or daily self-weighing (DSW) group. There were 3 testing visits: pre-holiday (v1: within 7d before Thanksgiving), post-holiday (v2: within 7d after New Year's Day), and a follow-up (v3: 14 weeks after v2). The DSW group were given Wi-Fi scales that provide graphical feedback of daily weight. They were instructed to perform DSW during the holidays and to try not to gain weight above baseline weights. Anthropometrics were measured at each visit.

ELIGIBILITY:
Inclusion Criteria:

* BMI of at least 18.5 kg/m2
* Recognizing or celebrating at least two holidays between November and January
* Access to WiFi

Exclusion Criteria:

* Current eating disorder, history of an eating disorder
* Involvement in a current weight loss and/or exercise program
* Pregnancy or nursing
* Any medications or chronic diseases affecting metabolism or body weight

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: jamie.cooper@uga.edu Cooper, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia - Department of Foods and Nutrition, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to share group averages through publication.

REFERENCES:
- [Derived] Kaviani S, vanDellen M, Cooper JA. Daily Self-Weighing to Prevent Holiday-Associated Weight Gain in Adults. Obesity (Silver Spring). 2019 Jun;27(6):908-916. doi: 10.1002/oby.22454. PMID 31119881

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Participants in this group received no intervention during the holiday season
Period: Overall Study
Arm/Group | Control | Daily Self-Weighing (DSW)
Started | 55 | 56
Completed | 53 | 51
Not Completed | 2 | 5
Not completed — Relocation | 2 | 4
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Daily Self-Weighing (DSW) | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (10.6) | 30.5 (12.1) | 29.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 14 | 15 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 56 | 111
Height [Mean (Standard Deviation); unit: cm] | 166.9 (9.5) | 167.5 (8.4) | 167.2 (9.0)
Weight [Mean (Standard Deviation); unit: kg] | 67.0 (13.1) | 66.6 (11.9) | 66.8 (12.5)
Total Body Fat Percentage [Mean (Standard Deviation); unit: percentage of body fat] | 25.9 (8.3) | 26.4 (6.7) | 26.2 (7.5)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 81.6 (11.2) | 79.3 (9.4) | 80.5 (10.3)
Hip Circumference [Mean (Standard Deviation); unit: cm] | 102.0 (8.6) | 101.4 (7.7) | 101.7 (8.2)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 115.2 (13.5) | 114.2 (11.4) | 114.7 (12.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 75.6 (9.2) | 73.3 (8.3) | 74.5 (8.8)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 172.4 (46.9) | 165.3 (32.0) | 168.9 (39.5)
Triglyceride [Mean (Standard Deviation); unit: mg/dL] | 79.8 (32.0) | 95.0 (51.5) | 87.4 (41.8)
HDL-Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 53.8 (11.7) | 50.9 (12.6) | 52.4 (12.2)
LDL-Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 102.7 (47.2) | 96.4 (24.6) | 99.6 (35.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — weight and height were combined to report BMI in kg/m^2
  kg/m^2 | 23.9 (3.5) | 23.6 (2.9) | 23.8 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (kg) From Pre- to Post-holiday and 14-week Follow-up Post-holiday
Description: Mechanical Beam Scale (Model 402KL, Health o Meter professional scales, McCook, IL, USA); Capacity: 390 lbs / 180 kg; Readability: 1/4 lb / 100 g.
Time Frame: Measured at 3 testing visits: Visit 1 (pre-holiday visit) occurred within 7 days before Thanksgiving, visit 2 (post-holiday visit) occurred within 7 days after New Year's Day, and visit 3 (follow-up visit) occurred 14 weeks after visit 2.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
kg
  Pre- to Post-Holiday | 2.65 (0.33) | -0.13 (0.27)
  Pre- to 14-week follow-up post-holiday | 1.51 (0.39) | -0.15 (0.35)

2. Secondary Outcome: Body Mass Index (BMI) (kg/m^2)
Description: weight and height will be combined to report BMI in kg/m^2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
kg/m^2
  Visit 2 | 24.9 (3.6) | 23.7 (2.9)
  Visit 3 | 24.5 (4.0) | 23.7 (2.9)

3. Secondary Outcome: Body Fat (%)
Description: Dual Energy X-Ray Absorptiometry
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of body fat
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
Percentage of body fat
  Visit 2 | 26.7 (8.5) | 25.3 (6.6)
  Visit 3 | 26.7 (8.3) | 26.1 (6.6)

4. Secondary Outcome: Waist Circumference (cm)
Description: Measuring tape
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
cm
  Visit 2 | 81.4 (10.8) | 80.6 (9.3)
  Visit 3 | 79.5 (10.5) | 79.1 (9.4)

5. Secondary Outcome: Hip Circumference (cm)
Description: Measuring tape
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
cm
  Visit 2 | 102.2 (10.0) | 102.2 (12.0)
  Visit 3 | 100.9 (9.9) | 100.1 (8.1)

6. Secondary Outcome: Concentration of Blood Triglyceride (mg/dL)
Description: Fasting blood draw
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
mg/dL
  Visit 2 | 81.6 (34.0) | 90.5 (54.3)
  Visit 3 | 80.3 (34.4) | 85.7 (39.7)

7. Secondary Outcome: Concentration of Blood High-density Lipoprotein (HDL) (mg/dL)
Description: Fasting blood draw
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
mg/dL
  Visit 2 | 52.1 (11.9) | 51.5 (15.3)
  Visit 3 | 53.0 (11.6) | 51.7 (13.2)

8. Secondary Outcome: Concentration of Blood Low-density Lipoprotein (LDL) (mg/dL)
Description: Fasting blood draw
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
mg/dL
  Visit 2 | 101.2 (49.6) | 91.3 (26.8)
  Visit 3 | 99.5 (50.0) | 90.0 (25.5)

9. Secondary Outcome: Concentration of Blood Total Cholesterol (TC) (mg/dL)
Description: Fasting blood draw
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Daily Self-Weighing (DSW)
Number analyzed (Participants) | 55 | 56
mg/dL
  Visit 2 | 169.6 (52.9) | 159.6 (34.6)
  Visit 3 | 168.6 (51.8) | 158.8 (39.7)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and other adverse events were not monitored/assessed.
Arm/Group | Control | Daily Self-Weighing (DSW)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03718000/Prot_SAP_000.pdf